CLINICAL TRIAL: NCT04517838
Title: Immune Response to Anti-HER2 Therapies
Brief Title: Immune Response to Anti-HER2 Therapies in Patients With HER2-Positive Stage I-IV Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC1937; NCI-2020-05781 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-011040 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Breast Adenocarcinoma; HER2-Positive Breast Carcinoma; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational Blood & Tissue Cohort: Patients with stage I-III disease undergo collection of blood samples at baseline, 8 and 16 weeks after starting treatment, and at the time of invasive disease recurrence. Patients with stage IV disease undergo collection of blood samples at baseline, 8 and 16 weeks after starting treatment, and at the time of progressive disease. Patients with stage IV disease with no disease progression ≥ 2 years on the same line of therapy undergo collection of blood samples at baseline, 8 and 16 weeks after starting treatment, and at the time of invasive disease recurrence. For all patients, tissue samples from previous biopsy and/or surgical resection are also collected on study.
  Interventions: Procedure: Biospecimen Collection
- Observational Tissue-Only Cohort: For patients with stage I-IV disease who received or previously completed anti-HER2 therapy, tissue samples from previous biopsy and/or surgical resection are collected on study.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and tumor tissue samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This study gathers information from the blood cells and tumor tissue during treatment with anti-HER2 therapies, such as trastuzumab, pertuzumab, lapatinib, or neratinib, in patients with HER2 positive stage I-IV breast cancer who are scheduled to start anti-HER2 therapy. The information gained from this study may help researchers better understand the relation between cell response and anti-HER2 therapies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES I. To determine the correlation between HER2 specific T-cell response in HER2-positive breast cancer patients with stage I-IV who receive anti-HER2 therapies, such as trastuzumab, pertuzumab, lapatinib, or neratinib and clinical responses.

II. To determine the correlation between antibody response in HER2-positive breast cancer patients with stage I-IV who receive anti-HER2 therapies, such as trastuzumab, pertuzumab, lapatinib, or neratinib and clinical responses.

III. To determine the correlation between host immune response in tumor tissue in HER2-positive breast cancer patients with stage I-IV who receive anti-HER2 therapies, such as trastuzumab, pertuzumab, lapatinib, or neratinib and clinical responses.

EXPLORATORY OBJECTIVES:

I. To estimate the proportion of patients who develop HER2-specific T cell and endogenous antibody responses.

II. To examine within individual patients trends in levels of HER2 CD4 T-cells, HER2 CD8 T-cells, and HER2-specific antibodies over the course of treatment.

III. To determine if combination therapy induces immunity to common breast cancer associated antigens (i.e. CEA, IGFBP2, and P53).

IV. To determine if induction of HER2-specific T cell or antibody immunity is associated with improved progression-free and overall survival in patients.

V. To determine if there are Fc gamma receptor (R) or HLA genotypes associated with the ability to generate immunity in response to anti-HER2 therapy.

VI. To determine whether anti-HER2 therapy induces HER2 loss and modulation of HER2-specific adaptive immune responses.

VII. To determine if loss-of-function mutations in antigen presenting genes are associated with recurrence in patients with HER2+ breast cancer.

VIII. To determine gene expression levels in tumors from patients who did not achieve pathologic complete response (pCR) that are associated with recurrence.

OUTLINE: This is an observational study. Patients are assigned to 1 of 2 cohorts.

BLOOD & TISSUE COHORT: Patients with stage I-III disease undergo collection of blood samples at baseline, 8 and 16 weeks after starting treatment, and at the time of invasive disease recurrence. Patients with stage IV disease undergo collection of blood samples at baseline, 8 and 16 weeks after starting treatment, and at the time of progressive disease. Patients with stage IV disease with no disease progression ≥ 2 years on the same line of therapy undergo collection of blood samples at baseline, 8 and 16 weeks after starting treatment, and at the time of invasive disease recurrence. For all patients, tissue samples from previous biopsy and/or surgical resection are also collected on study.

TISSUE-ONLY COHORT: For patients with stage I-IV disease who received or previously completed anti-HER2 therapy, tissue samples from previous biopsy and/or surgical resection are collected on study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological confirmed adenocarcinoma of the breast stage I-IV from the American Joint Committee on Cancer staging 8th edition
* Any estrogen receptor (ER) or progesterone receptor (PR) but HER2 positive defined as per the most current American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guideline
* Provide written informed consent
* Willingness to provide blood samples for correlative research purposes
* BLOOD AND TISSUE COHORT: Scheduled to start new anti-HER2 therapy/therapies
* TISSUE-ONLY COHORT: Received or previously completed anti-HER2 therapy/therapies

Exclusion Criteria:

* Immunocompromised patients including patients known to be human immunodeficiency virus (HIV) positive
* Receiving systemic steroid therapy or any other immunosuppressive therapy =< 30 days prior to registration. NOTE: Inhaled steroids, low-dose corticosteroids (e.g. equivalent to or less than oral prednisone 10 mg daily), and steroid use for primary prevention of nausea per institutional guidelines are allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage I-IV HER2 positive breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2020-07-31 (Actual); Primary Completion 2028-07-27 (Estimated); Study Completion 2028-07-27 (Estimated)

PRIMARY OUTCOMES:
HER2 specific T-cell response and clinical response | Up to 16 weeks
  Defined as (1) a 2-fold or greater increase in HER2-specific T cells or HER2-specific antibodies at any point during treatment if pre-treatment levels of HER2-specific T cells or antibodies are detectable, or (2) HER2-specific T cells or HER2-specific antibodies at any point during treatment if pretreatment levels of HER-2 binding activity are non-detectable.
Antibody response and clinical response | Up to 16 weeks
  Defined as (1) a 2-fold or greater increase in HER2-specific T cells or HER2-specific antibodies at any point during treatment if pre-treatment levels of HER2-specific T cells or antibodies are detectable, or (2) HER2-specific T cells or HER2-specific antibodies at any point during treatment if pretreatment levels of HER-2 binding activity are non-detectable.

OTHER OUTCOMES:
Proportion of patients who develop HER2-specific T cell and endogenous antibody responses | Up to 16 weeks
  A two sided alpha=0.10 test of proportions will be used to assess whether the proportion of women who develop a HER2-specific immune response differs between the women who develop a tumor response and those who do not.
Levels of HER2 CD4 T-cells, HER2 CD8 T-cells, and HER2-specific antibodies | Up to 16 weeks
  Descriptive statistics will be used to quantify T cell or antibody response within each cohort of patients, namely (neo)adjuvant vs. metastatic setting and within each anti-HER2 treatments (i.e. trastuzumab, pertuzumab, lapatinib, or neratinib).
Association between combination therapy and immunity to common breast cancer associated antigens | Up to 16 weeks
  Descriptive statistics will be used.
Association between HER2-specific T cell or antibody immunity and improved progression-free survival | Up to 16 weeks
  Descriptive statistics will be used.
Association between HER2-specific T cell or antibody immunity and improved overall survival in patients | Up to 16 weeks
  Descriptive statistics will be used.
Association between anti-HER2 therapy and HER2 loss and modulation of HER2-specific adaptive immune responses | Up to 16 weeks
  Descriptive statistics will be used.
Association between loss-of-function mutations and recurrence | Up to 16 weeks or recurrence
  Descriptive statistics will be used.
Association between gene expression levels and recurrence | Up to 16 weeks or recurrence
  Descriptive statistics will be used.
Association between Fc gamma receptor (R) or human leukocyte antigen (HLA) genotypes and ability to generate immunity | Up to 16 weeks
  Descriptive statistics will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Saranya Chumsri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials